CLINICAL TRIAL: NCT01861704
Title: Post-market Study to Capture Information Regarding Performance of Extended Wear Hearing Aid Lyric2 Compared to Lyric
Brief Title: Post-market Study to Capture Information Regarding Performance of Lyric2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 000.000.004.858
Record Dates: First submitted 2013-03-21; First posted 2013-05-24 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Hearing Loss
Keywords: Mild to moderate hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyric (Active Comparator): Silver Lyric device
  Interventions: Device: Lyric
- Lyric2 (Active Comparator): Lyric2 (Barracuda) device
  Interventions: Device: Lyric2

INTERVENTIONS:
Device: Lyric — Extended wear hearing instrument
  Arms: Lyric
Device: Lyric2 — Extended wear hearing instrument
  Arms: Lyric2

SUMMARY:
Randomized post market study comparing Lyric to Lyric2 capturing information regarding comparative performance and safety.

DETAILED DESCRIPTION:
Randomized post market study comparing extended wear hearing aids Lyric to Lyric2 capturing information regarding comparative performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90 years at the time of enrollment in the study
* Mild to moderately-severe hearing loss bilaterally, or unilaterally if normal hearing in other ear
* Fluent in English
* Willingness to comply with all study requirements

Exclusion Criteria:

* Scuba dives or sky dives
* Underwater swimming or dives into the water
* Handicaps that would restrict participation in all the evaluations
* Hearing loss of neural or central origin
* Unrealistic expectations regarding benefits and limitations inherent in the devices
* Chemotherapy within the last six months
* Compromised immune system
* Radiation to head or neck
* Perforated tympanic membrane
* History of cholesteatoma
* Active outer or middle ear pathology
* High levels of anticoagulant therapy
* Insulin-dependent and/or uncontrolled diabetes
* Contact dermatitis
* Bleeding disorder
* Unwillingness or inability to comply with all study requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Arbogast, Principal Investigator — Employee
Locations (1):
- InSound Medical, Newark, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients are fitted according to their ear size and experience level. Patients with a different experience level for each ear are only counted once.
Groups:
- Lyric2: Lyric2 (Barracuda) device
  Lyric: Extended wear hearing instrument
Period: Overall Study
Arm/Group | Lyric | Lyric2
Started | 70 | 107
Completed | 67 | 104
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyric | Lyric2 | Total
Number analyzed (Participants) | 70 | 107 | 177
Age, Customized [Number; unit: participants]
  <=18 years of age | 0 | 0 | 0
  >18 years of age | 70 | 107 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 35 | 48
  Male | 57 | 72 | 129
Region of Enrollment [Number; unit: participants]
  United States | 70 | 107 | 177

OUTCOME MEASURES:

1. Primary Outcome: Immediate Refit Upon Device Removal
Description: Upon device removal, a qualified audiologist examined subjects' ears to evaluate their availability to be immediately refit with another hearing aid device. It is not uncommon for patients being fitted with these types of devices to experience slight irritation on an initial experience with the device. In particular, those being fit with the Lyric or Lyric2.0 for the first time first undergo the device sizing process, which slightly increases stress on the ear.
Time Frame: Following device removal at the same appointment (Up to 24 hours after removal)
Population: Only ears from experienced users were taken into account, i.e. only users that have previously worn an extended wear device. Some patients previously worn only one hearing instrument, therefor a significant number of patients were only fitted with one instrument
Measure: Number (90% Confidence Interval); unit: percentage of ears
Units Other Than Participants: Experienced ears
Groups:
- Lyric: Silver Lyric device
  Lyric: Extended wear hearing instrument
  Only experienced ears counted
- Lyric2: Lyric2 (Barracuda) device
  Lyric: Extended wear hearing instrument
  Only experienced ears counted
Arm/Group | Lyric | Lyric2
Number analyzed (Participants) | 35 | 41
Number analyzed (Experienced ears) | 65 | 61
percentage of ears | 78 [68 to 86] | 93 [86 to 98]

2. Secondary Outcome: Device Comfort
Time Frame: During useful lifespan of device
Reporting Status: Not Posted

3. Secondary Outcome: Gain, Speech Understanding and Sound Quality
Time Frame: During useful lifespan of device
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lyric | Lyric2
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/107
Other Adverse Events (participants affected / at risk) | 4/70 | 6/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyric (N=70) | Lyric2 (N=107)
Sound Quality -> Fine tuning (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Complaint in follow up or on the phone No removal, only fine tuning the settings
Acoustic Feedback -> Removal (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Complaint in follow up or on the phone, device got removed
Discomfort / Pain -> Removal (Ear and labyrinth disorders) | 1 (1) | 2 (2) — Complaint in follow up or on the phone, device got removed
Handling -> Removal (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Handling issues, patient removed the device himself not knowing that it cannot be reinserted
Sound Quality -> Removal (Ear and labyrinth disorders) | 0 (0) | 2 (2) — Sound quality issues with the device leading to a removal and exchange of the hearing aid
Handling -> Fine tuning (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Issue with handling of the device that could be resolved by retraining the patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes